CLINICAL TRIAL: NCT03145831
Title: An Open-Label, Long-Term Safety Study of Long-acting Human Growth Hormone Somavaratan (VRS-317) in Japanese Children With Growth Hormone Deficiency
Brief Title: A Long-Term Safety Study of Somavaratan in Japanese Children With Growth Hormone Deficiency
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The primary endpoint of non-inferiority to daily therapy in the pediatric Phase 3 study was not achieved
Sponsor: Versartis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J15VR6
Record Dates: First submitted 2017-04-05; First posted 2017-05-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Growth Hormone Deficiency
Keywords: Pediatrics
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Somavaratan (Experimental): fusion protein, subcutaneous bolus injection, 3.5 mg/kg twice monthly
  Interventions: Drug: Somavaratan

INTERVENTIONS:
Drug: Somavaratan — All subjects will receive somavaratan 3.5 mg/kg twice monthly (every 15 days ± 2 days). Administered as a subcutaneous bolus injection.
  Other Names: VRS 317

SUMMARY:
This study is a multi-center, open-label safety study assessing long-term somavaratan administration.

DETAILED DESCRIPTION:
This study is a multi-center, open-label safety study assessing long-term somavaratan administration. It is open to subjects completing a somavaratan Japanese Phase 2/3 study (Protocol J14VR5) in children with growth hormone deficiency (GHD), as well as approximately 20 new children currently receiving daily rhGH therapy for GHD (switch subjects). For switch subjects, the first dose of somavaratan will be administered approximately 48 hours after the last dose of the daily rhGH. All subjects will receive somavaratan 3.5mg/kg twice-monthly. The study will be conducted at approximately 40 medical institutions in Japan.

ELIGIBILITY:
Inclusion Criteria:

1. Chronological Age ≥ 3.0 years.
2. Pre-pubertal status: Absent breast development in girls, testicular volume < 4.0 mL in boys.
3. Subjects with GHD (diagnosed according to the current diagnostic guidelines) who are receiving treatment with daily rhGH.
4. Normal thyroid function at screening visit in subjects not being treated for hypothyroidism. Subjects requiring thyroxine replacement must be considered adequately treated by the PI and Medical Monitor.
5. Normal adrenal function (morning cortisol and/or local stimulation test) at screening visit or within 6 months of the screening visit, in subjects not being treated for adrenal insufficiency. Subjects with adrenal insufficiency must receive glucocorticoid treatment for a minimum of 4 weeks before study drug administration.
6. Pathology relating to cause of GHD must be stable for at least 6 months prior to screening.
7. Willingness to discontinue daily rhGH therapy.
8. Legally authorized representatives must be willing and able to give informed consent

Exclusion Criteria:

* 1. Prior (in the last 12 months) or concomitant treatment with a growth promoting agent other than rhGH [e.g., IGF-I, GH releasing hormone (GHRH), sex steroids (except when used as primer for GH stimulation test), aromatase inhibitors and/or GnRH agonist].

  2. Current significant disease (e.g., diabetes, cystic fibrosis, renal insufficiency). In all cases of concurrent disease, screening must be approved in writing by the medical monitor.

  3. Chromosomal aneuploidy, significant gene mutations (other than those that cause GHD) or confirmed diagnosis of a named syndrome (e.g., Russell Silver, Prader Willi, Turner, etc.).

  4. Birth weight and/or birth length less than 5th percentile for gestational age using local gestational age growth charts.

  5. Prolonged daily (> 14 days) use of anti-inflammatory doses of oral glucocorticoids.

  6. Prior history of malignancy. 7. Treatment with an investigational drug in the 30 days prior to screening. 8. Known allergy to constituents of the study drug formulation. 9. Ocular findings suggestive of increased intracranial pressure and/or retinopathy at screening.

  10. Significant spinal abnormalities including scoliosis, kyphosis, Chiari malformation, and spina bifida variants.

  11. Significant abnormality in screening laboratory studies (as assessed by PI and medical monitor).

  12. Current social conditions which would prevent completion of study activities (e.g., planned family move to a distant location).

  13. History of pancreatitis or undiagnosed chronic abdominal pain. 14. History of spinal or total body irradiation. 15. Presence of other pituitary hormone deficiencies that are not properly treated.

  16. Unwillingness to provide consent for participation in all trial activities

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 12 months
  Incidence and severity of adverse events

SECONDARY OUTCOMES:
Height velocity | 12 months
  Comparison of Height Velocity (HV) and HV-SDS before and after switching therapy
IGF-I expression | 12 months
  Change from Day 1
Immunogenicity | 12 months
  Evaluated by anti-drug antibody response

CONTACTS AND LOCATIONS:
Overall Officials: Will Charlton, MD, Study Director — Vesrartis
Locations (1):
- Eric Humphriss, Menlo Park, California, United States

IPD SHARING:
Plan to Share IPD: No